CLINICAL TRIAL: NCT01924910
Title: A Single Wintertime Dose of Vitamin D3 to Prevent Winter Decline in Vitamin D Concentrations in Healthy Adults: A Pilot Study
Brief Title: A Single Wintertime Dose of Vitamin D3 to Prevent Winter Decline in Vitamin D Status in Healthy Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Vin Tangpricha, MD, PH.D, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00061103; OnceYearlyD (Other: Other)
Record Dates: First submitted 2013-08-12; First posted 2013-08-19 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Vitamin D Deficiency
Keywords: Healthy, by self report
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol; Single Person

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Pill (Placebo Comparator): Received identical pills that do not contain vitamin D. Blood levels of 25(OH)D determined at 10 days, 3 months, and 1 year following placebo dose.
  Interventions: Dietary Supplement: Placebo
- Vitamin D (Active Comparator): 250,000 IU cholecalciferol as single, oral dose. Blood levels 25(OH)D measured at 10 days, 3 months, and 1 year following dose.
  Interventions: Dietary Supplement: 250,000 IU cholecalciferol as single, oral dose

INTERVENTIONS:
Dietary Supplement: 250,000 IU cholecalciferol as single, oral dose — 250,000 IU cholecalciferol (vitamin D3) provided as a single oral dose.
  Other Names: vitamin D3
  Arms: Vitamin D
Dietary Supplement: Placebo
  Arms: Placebo Pill

SUMMARY:
The purpose of this study is to determine if a single dose of vitamin D administered orally in the fall will provide adequate vitamin D in healthy individuals for the duration of the winter, during which vitamin D levels are known to decrease. The investigators are also interested in finding out if this level of vitamin D will provide adequate levels for the remainder of the year. While the benefits of once-yearly vitamin D administration are clear for patients with osteoporosis, osteomalacia, rickets, and other conditions associated with vitamin D deficiency and high bone turn-over, studies have not been performed in which high doses of vitamin D were used to prevent the seasonal decline of vitamin D concentrations in healthy individuals. These findings could provide evidence to support vitamin D administration to healthy individuals in the wintertime to improve health outcomes, and provide the basis for additional studies in both healthy and sick populations.

DETAILED DESCRIPTION:
Vitamin D, synthesized from 7-dehydrocholesterol during ultraviolet- B exposure, aids in the absorption of calcium from the G.I. tract. Indirectly, by maintaining optimal calcium homeostasis, adequate vitamin D concentrations are essential in skeletal health (by preventing rickets and osteomalacia), cardiovascular health (by lowering the risk for hypertension), and ultimately decreasing mortality. Due to decreased direct sunlight exposures in the winter (characterized by limited outdoor activity, increased clothing coverage, and angle of the sun), vitamin D concentrations are shown to decline in individuals over the winter. Once-yearly administration of a bolus of vitamin D offers a means of preventing the seasonal decline in vitamin D status and preventing vitamin D deficiency. If proven successful, a once-yearly dose of vitamin D would provide improved compliance relative to daily or monthly dosing and provide an inexpensive and easy way to ensure optimal concentrations of vitamin D year-round.

This pilot study plans to investigate if once a year dosing with vitamin D during the winter months in self-identified healthy adults will be effective in maintaining optimal vitamin D status for the entire year. In brief, this study will be a randomized, double blind, placebo-controlled study to evaluate the efficacy of 250,000 IU of vitamin D3 compared to placebo given once in 30 healthy individuals (15 subjects per arm) in November. The serum 25(OH)D (the best measurable level of vitamin D status) will be measured after both 3-4 months and 1 year to determine the efficacy of the dose relative to the 15 healthy controls. The intent of this clinical investigation is not to evaluate the dietary supplement's ability to diagnose, cure, mitigate or prevent disease. This study is to evaluate blood concentrations of this regimen of vitamin D.

Ultimately, this study hopes to determine if a single dose of vitamin D administered orally in the fall will provide adequate vitamin D in healthy young individuals for the 3 months during winter, during which vitamin D levels are known to decrease, and over the entire year. These findings could provide evidence to support vitamin D administration to healthy individuals in wintertime to improve health outcomes, and provide the basis for additional studies in both healthy and sick populations.

Secondary outcomes of this study will evaluate other hypothesized effects of vitamin D on biomarkers affecting health status and immunity, including markers of inflammation and markers of iron status.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult (by self-report) between ages 18-65

Exclusion Criteria:

1. reported granulomatous conditions
2. history of kidney disease (renal failure, renal stones, serum creatinine over 0.06 ng/mL in the past)
3. diabetes
4. currently taking anticonvulsants, barbituates, antihypertensives, steroids of any form, or drugs that effect bone metabolism
5. history of calcium or bone abnormalities (including osteoporosis)
6. primary hyperparathyroidism
7. thyrotoxicosis
8. Paget's disease
9. history of malignancy
10. known liver disease
11. calcium supplements >1000 mg/day
12. complete immobilization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
blood levels of 25(OH)D | 3 months
  Measure blood levels of 25(OH)D, an indicator of vitamin D status, at 10 days, 3 months, and 1 year following vitamin D or placebo dose.

SECONDARY OUTCOMES:
Blood Calcium level | 10 days
  Measured blood calcium levels at 10 days following dose. This measure assessed safety of large vitamin D dose regarding its potential to cause hypercalcemia.
Blood pro-inflammatory cytokines | baseline, 10 days, 3 months, 1 year
  Measured blood cytokine (IL-6, IL-1B, IL-8, MCP-1) concentrations at baseline, 10 days, 3 months, and 1 year
Blood hepcidin concentration | baseline, 10 days
  Measured blood hepcidin concentrations at baseline and 10 days
Blood markers of iron status | baseline, 10 days
  Measured blood ferritin concentrations at baseline and 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Vin Tangpricha, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University Campus, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Kearns MD, Binongo JN, Watson D, Alvarez JA, Lodin D, Ziegler TR, Tangpricha V. The effect of a single, large bolus of vitamin D in healthy adults over the winter and following year: a randomized, double-blind, placebo-controlled trial. Eur J Clin Nutr. 2015 Feb;69(2):193-7. doi: 10.1038/ejcn.2014.209. Epub 2014 Oct 1. PMID 25271011